CLINICAL TRIAL: NCT05946226
Title: A Phase I, Open-label, Multi-center, Dose-escalation Study to Evaluate the Safety, Feasibility, and Preliminary Efficacy of IMC002 in Patients With Claudin18.2-positive Advanced Digestive System Tumors
Brief Title: A Phase I Trial to Evaluate the Safety of IMC002 in Advanced Digestive System Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Immunofoco Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC002-RT01
Record Dates: First submitted 2023-06-15; First posted 2023-07-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Advanced Digestive System Tumor

STUDY DESIGN:
Intervention Model Description: A classic 3+3 model will be used to dose escalation 3 doses will be used: 1×10^8, 2.5×10^8 and 5×10^8 CAR-T cells/ patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMC002 dose 1-3 (Experimental): IMC002 single infusion
  Interventions: Biological: IMC002 injection

INTERVENTIONS:
Biological: IMC002 injection — three different IMC002 Doses will be escalated in "3+3" design
  Other Names: Autologous Claudin 18.2 specific CAR-T cell injection

SUMMARY:
This is an open-label, multi-center, dose-escalation clinical study to evaluate the safety, feasibility, and preliminary efficacy of IMC002 in patients with CLDN18.2 positive digestive system tumors including but not limited to advanced gastric cancer, esophagogastric junction adenocarcinoma, and advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation clinical study to evaluate the safety, feasibility, and preliminary efficacy of IMC002 in patients with CLDN18.2 positive digestive system tumors including but not limited to advanced gastric cancer, esophagogastric junction adenocarcinoma, and advanced pancreatic cancer.

Approximately 9-18 patients with CLDN18.2-positive advanced digestive system tumors will be sequentially enrolled into 3 dose escalation cohorts to evaluate the safety and feasibility of autologous IMC002 treatment. Following enrolment, patients will undergo leukapheresis and IMC002 product preparation. Patients may receive bridging therapies if the disease progresses rapidly as determined by the investigator. After treatment with cyclophosphamide, fludarabine and nab-paclitaxel lymphodepletion, patients will be assigned to one of three dose escalation cohorts 1.0×108, 2.5×108, or 5.0×108 CAR-T cells. All patients will be given a single dose of IMC002 infusion. All patients will be followed as inpatient for 14 days. When all patients of a cohort have been observed for 28 days and no DLT criteria have been met, patients will be enrolled in next higher dose cohort. All enrolled patients will follow the same study treatment schedule and procedural requirements.

This study is divided into a screening period, a lymphodepleting (LD) chemotherapy period, a treatment period, a primary follow-up period up to 12 weeks and a long-term follow-up period for up to 15 years post infusion.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures
* Age > 18 and ≤70 years
* Patients with histologically or cytologically confirmed locally advanced/metastatic digestive system tumors including but not limited to advanced gastric cancer at least failed two lines of SOC, esophagogastric junction adenocarcinoma, and advanced pancreatic cancer failed at least one line SOC;
* Must have CLDN18.2 positive tumor expression histologically as determined by IHC (defined as positive rate of tumor cells≥40% and staining intensity ≥2+ ) or a biopsy if archived tumor sample is not available; representative tumor samples (primary or metastatic, archived or newly collected) are expected to be obtained
* Expected survival time ≥12 weeks
* Measurable or evaluable disease per RECIST1.1
* ECOG performance status score of 0-1
* Adequate organ and bone marrow function. If any laboratory test results are abnormal with reference to the criteria below, a repeat test can be performed within 1 week. If the test results are still abnormal, the patient fails screening.
* Recovery to grade 0-1 from AEs related to prior anticancer therapy or to an acceptable level for inclusion/exclusion criteria except alopecia and vitiligo
* Female of childbearing age must undergo a serum pregnancy test with negative results at screening and infusion; Female of childbearing age or male patients whose sexual partners are females of childbearing age are willing to take medically approved high-efficiency contraceptive measures such as intrauterine devices or condoms from the time of signing the informed consent to 1 year after infusion (women of childbearing age include premenopausal women and women within 24 months of post menopause).

Exclusion Criteria:

* Pregnant and lactating women
* Human immunodeficiency virus (HIV) antibody positive; acute or chronic active hepatitis B; acute or chronic active hepatitis C Hepatitis. Syphilis antibody positive; cytomegalovirus (CMV) infection; Epstein-Barr (EB) virus infection.
* Active or clinically poorly controlled serious infections
* Uncontrollable pleural effusion, pericardial effusion and ascites effusion existed before enrollment.
* Extensive or diffuse lung or liver metastases
* Oxygen saturation ≤95% without oxygen inhalation
* With other diseases that may limit their participation in this study, such as pulmonary embolism, chronic obstructive pulmonary disease, symptomatic or poorly controlled interstitial lung disease, or clinically significant abnormal lung function tests
* Known prior or current hepatic encephalopathy requiring treatment; patients with current or history of central nervous system (CNS) disease. Autoimmune diseases; CNS metastases or meningeal metastases with clinical symptoms, or other evidence that the patient's CNS or meningeal metastases have not been controlled, and are judged not suitable for the study by the investigator
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure > 100 mmHg after standardized antihypertensive drug treatment); not well controlled diabetes mellitus [fasting plasma glucose (FPG) ≥10.2mmol/L].
* Presence of any of clinical cardiac symptoms or disorders
* Evidence of major coagulopathy or other significant bleeding risk
* Systemic steroids equivalent to >15mg/day prednisone within 2 weeks before leukapheresis, except inhaled or topic steroids
* Requiring systemic therapy with corticosteroids or other immunosuppressive drugs during the treatment period. Presence of any active autoimmune disease, or history of autoimmune disease expect recur.
* Previous or concomitant other malignancies
* Have received other gene therapies including but not limited to any CAR-T and TCR-T therapy
* Anti-tumor therapies other than for the pretreatment and bridging therapies < 5 half-lives or 28 days (whichever is shorter) prior to study treatment
* Any investigational drugs or study drugs from a previous clinical study within 30 days prior to signing the informed consent; traditional Chinese medicine with anti-tumor activities within 2 weeks prior to the study treatment
* History of serious allergic disease or known allergy to any component of the study treatments
* With severe mental disorders
* Any issue that would impair the ability of the patient to receive or tolerate the planned treatment, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicity (DLTs) within 28 days after IMC002 infusion | within 28 days
  safety profile

SECONDARY OUTCOMES:
ORR after IMC002 infusion | upto 96 weeks
  efficacy endpoints
Incidences and severity of treatment-related adverse events (TRAEs) | upto 96 weeks
  AEs
cytokine levels in the blood | upto 96 weeks
  IL-6, TNF-α, IL-10, IL-2, IFN-γ and other cytokines in peripheral
CAR-positive cell counts in peripheral blood | upto 96 weeks
  Cmax

OTHER OUTCOMES:
Immunogenicity parameters in peripheral blood | upto 96 weeks
  Number of Participants with presence of human anti-CAR antibodies (ADA)
long-term safety | upto 96 weeks
  Number of Participants with presence of RCL in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, Pro., Principal Investigator — Chinese PLA General Hospital
Locations (7):
- China (7):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Shandong Cancer Hospital, Jinan, Shandong
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No